CLINICAL TRIAL: NCT02865447
Title: A Dual Energy X-ray Absorptiometry (DXA) Evaluation of Bone Density Changes After Hip Replacement. Performance of the PROFEMUR® PRESERVE Hip Stem in Total Hip Arthroplasty, Two-Year Clinical and DXA Analysis
Brief Title: Evaluation of Bone Mineral Density Changes After Total Hip Replacement: A Two-Year Clinical and DXA Analysis
Status: Completed | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Collaborators: Orthopaedic Specialty Clinic of Spokane, PLLC (Other)
Responsible Party: Sponsor
Other Study IDs: 15-LJH-001
Record Dates: First submitted 2016-07-01; First posted 2016-08-12 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Joint Disease
Keywords: dual energy x-ray absorptiometry; DEXA; DXA; total hip arthroplasty; PROFEMUR; PRESERVE; bone mineral density; BMD; osteoarthritis; THA; musculoskeletal disease
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Musculoskeletal Diseases | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PRESERVE total hip arthroplasty implant: Subjects to be prospectively implanted with the PROFEMUR PRESERVE total hip arthroplasty implant
  Interventions: Device: total hip arthroplasty implant

INTERVENTIONS:
Device: total hip arthroplasty implant — PROFEMUR PRESERVE total hip arthroplasty femoral stem
  Other Names: PROFEMUR PRESERVE

SUMMARY:
Sponsor is conducting this post-market study to evaluate the clinical outcome and femoral bone mineral density (BMD) changes associated with the PROFEMUR® PRESERVE hip stem when used as indicated for primary total hip arthroplasty in patients with osteoarthritis of the hip joint.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, subjects must meet all of the following criteria:

* Subject is minimum age 21 years, maximum age of 80
* Subject is a candidate for primary THA for osteoarthritis of the hip
* Subject is able to undergo primary elective THA procedure
* Subject is willing and able to complete required study visits and assessments
* Subject is willing to sign the Institutional Review Board/Ethics Committee (IRB/EC) approved Informed Consent document.

Exclusion Criteria:

Subjects will be excluded if they meet any of the following criteria:

* Overt infection;
* Distant foci of infections (which may cause hematogenous spread to the implant site);
* Rapid disease progression as manifested by joint destruction or bone absorption apparent on roentgenogram;
* Skeletally immature (less than 21 years of age at time of surgery);
* Inadequate neuromuscular status (e.g., prior paralysis, fusion, and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable;
* Neuropathic joints;
* Known Hepatitis or HIV infection;
* Neurological or musculoskeletal disease that may adversely affect gait or weight-bearing
* Subjects with known osteoporosis of the affected hip
* Subjects with prior arthroplasty of the affected hip
* Subjects that are clinically obese (>40 body mass index [BMI])
* Subjects with femoral dysplasia of the affected hip
* Subjects with trochanteric osteotomy of the affected hip
* Subject with inflammatory arthritis of the affected hip
* Subjects currently taking, or have taken within 12 months of enrollment, bisphosphonates, parathyroid hormone (PTH), fluoride therapy or strontium ranelate or patients taking other chronic medications that in the investigator's opinion are known to affect BMD in a substantial way
* Subjects with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Subjects currently enrolled in another clinical study which could affect the endpoints of this protocol
* Subjects with known substance abuse issues
* Subjects who are incarcerated or have pending incarceration

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the investigator's private orthopedic practice from among patients who require a total hip arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral density (BMD), per dual energy x-ray absorptiometry (DXA) imaging, from standard and custom Gruen zones around the femoral stem. | 1 week Postoperative, 6 weeks, 6 Months, 12 Months, and 24 Months Postoperative

SECONDARY OUTCOMES:
Hip functional outcomes will be assessed using the Harris Hip score. | Preoperative, 6 weeks Postoperative, 6 Months, 12 Months, and 24 Months Postoperative
Implant loosening will be assessed by the presence of radiographic lucencies around the femoral stem. | 6 weeks Postoperative, 6 Months, 12 Months, and 24 Months Postoperative
Implant survivorship of the femoral stem will be calculated. | 1 week Postoperative, 6 weeks, 6 Months, 12 Months, and 24 Months Postoperative
Rate of complications will be assessed. | Preoperative, 6 weeks Postoperative, 6 Months, 12 Months, and 24 Months Postoperative
Hip functional outcomes will be assessed using the Forgotten Joint Score. | 6 weeks Postoperative, 6 Months, 12 Months, and 24 Months Postoperative

CONTACTS AND LOCATIONS:
Overall Officials: David Scott, MD, Principal Investigator — Spokane Joint Replacement Center, Inc.
Locations (1):
- Spokane Joint Replacement Center, Spokane, Washington, United States